CLINICAL TRIAL: NCT04375761
Title: Human Epidemiology and Response to SARS-CoV-2 (DAIT-COVID-19-001)
Brief Title: COVID-19: Human Epidemiology and Response to SARS-CoV-2
Acronym: HEROS
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: DAIT-COVID-19-001
Record Dates: First submitted 2020-04-30; First posted 2020-05-05 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Coronavirus Disease 2019 (COVID-19); SARS-CoV-2
Keywords: COVID-19; SARS-CoV-2; Public Health Surveillance; Participants in NIH-funded studies (and their families)
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal, peripheral blood and stool samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SARS-CoV-2 Surveillance: Total Group: Participants either currently or in the past, enrolled in National Institutes of Health (NIH)-funded cohort studies, and their families (household contacts).
  Active surveillance for detection of SARS-CoV-2 for 6 months, beginning with enrollment. During surveillance, biological samples will be collected by the family at established intervals and symptom and exposure surveys will be completed at the time that biological samples are collected.
  Interventions: Procedure: Collection of Biological Samples; Procedure: Symptom and Exposure Surveys

INTERVENTIONS:
Procedure: Collection of Biological Samples — Biological samples will be collected throughout the study at regular intervals (every 2 weeks) in addition to when illness event(s) occur. All biological samples (e.g. nasal swabs, peripheral blood, stool) will be collected by the caregiver at home using materials provided to the family. At the end of study, additional samples (e.g. nasal secretion and/or saliva samples) may be collected by the family or study staff at a site visit, if feasible.
Procedure: Symptom and Exposure Surveys — Symptom and exposure surveys (questionnaires) will be completed throughout the study at regular intervals (every 2 weeks) in addition to when illness event(s) occur. The primary household contact/caregiver will be the designee for ensuring timely questionnaires completion and submission for all household study participants.
  Other Names: Symptom and Exposure Questionnaires

SUMMARY:
The human disease caused by SARS-CoV-2 is called COVID-19. In most cases, COVID-19 presents as a mild to moderate respiratory illness. But it can also be more severe and even lead to death.

The purpose of this study is to:

* Determine the prevalence of SARS-CoV-2 carrier status over time in children and parents
* Determine the prevalence of antibody development over time in children and parents
* Compare carrier status and antibody development for children with asthma and/or other atopic conditions (e.g. eczema) versus children without asthma and/or other atopic conditions
* Investigate the presence of SARS-CoV-2 exposure in historical samples from enrolled participants

DETAILED DESCRIPTION:
The study population will include children that are participants in NIH-funded cohort studies and their families (household contacts).The intent is to recruit families that have experience with the collection of respiratory samples.

The objective of this surveillance study is to identify the rate of infection in children and what, if any effect, atopy has on the SARS-CoV-2 carrier status.

The initial surveillance interval for participants will be 6 months and, depending upon the findings, may be extended. During surveillance, biological samples will be collected by the family at established intervals and symptom and exposure surveys will be completed remotely via a smart phone, on-line, or phone communications at the time the biological samples are collected.

ELIGIBILITY:
Inclusion Criteria:

Household members who meet all of the following criteria are eligible for enrollment as study participants:

* The index participant, defined as an individual who either is or has been a participant in an NIH-funded clinical research study from which information on respiratory conditions, including asthma, and other atopic and allergic diseases is available, is:

  * ≤21 years of age, and
  * Lives with caregiver(s).
* The index participant and/or caregiver understands the study procedures and is willing to conduct these procedures at home;
* Have the ability to use either a computer or a smart phone to link to and respond to the study questionnaires:

  --Exception: When the family is willing to speak with a study member to answer the questionnaires in the event of not having access to a computer or a smart phone.
* The index participant and caregiver will reside in the United States, including Puerto Rico, for the duration of the study;
* The index participant will live with the caregiver for at least 50% of the time for the duration of the study;
* An English or Spanish speaker is available to:

  * Serve as the primary contact, and
  * As the person who will be responsible for the completion of questionnaires and the collection of study biological samples; and,
* To participate as a sibling (of the index participant), must be under 21 years of age and live in the same home as the index participant and caregiver.

Exclusion Criteria:

-Past or current medical problems, which, in the opinion of the site investigator may:

* Pose risks from participation in the study
* Interfere with the participant's ability to comply with study requirements, or
* Impact the quality or interpretation of the data obtained from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: NIH-funded study participants (index participants) and their families This includes participants who have asthma and/or other atopic or allergic conditions, as well as healthy index participants, all with extensive medical information and information on atopic and allergic status available as a result of their participation in an NIH-funded study. As many of these are birth cohort studies, there is extensive information available on the parents. The majority of the families have experience with collection of respiratory samples and completing respiratory questionnaires.
Sampling Method: Probability Sample
Enrollment: 5599 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina V. Hartert, MD, MPH, Study Chair — Vanderbilt University School of Medicine, Dept. of Medicine
Locations (20):
- United States (20):
  - Children's Hospital Colorado: Inner City Asthma Consortium (ICAC) Site, Aurora, Colorado
  - Children's Hospital Colorado: Outcome Measures in Eosinophilic Gastrointestinal Disorders Across the Ages (OMEGA) Site, Aurora, Colorado
  - Children's National Medical Center: Inner City Asthma Consortium (ICAC) Site, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago: Food Allergy Outcomes Related to White and African American Racial Differences (FORWARD) and Improving Technology-Assisted Recording of Asthma Control in Children (iTRACC) Site, Chicago, Illinois
  - Massachusetts General Hospital:Childhood Microbiome (CHIME) and Wheezing Index (WIND) Site, Boston, Massachusetts
  - Boston Children's Hospital: School Inner-City Asthma Study (SICAS-2), Environmental Assessment of Sleep in Youth (EASY), Severe Asthma Research Program (SARP) and Preventing Asthma in High Risk Kids (PARK) Site, Boston, Massachusetts
  - Boston Medical Center: Inner City Asthma Consortium (ICAC) Site, Boston, Massachusetts
  - Henry Ford Health System: Childhood Allergy Study (CAS) Site, Detroit, Michigan
  - Henry Ford Health System: Inner City Asthma Consortium (ICAC) Site, Detroit, Michigan
  - Henry Ford Health System: Microbes, Asthma, Allergy and Pets (MAAP) and Wayne County Health, Environment, Allergy, and Asthma Longitudinal Study (WHEALS) Site, Detroit, Michigan
  - St. Louis Children's Hospital: Inner City Asthma Consortium (ICAC) Site, St Louis, Missouri
  - Columbia University Medical Center: Inner City Asthma Consortium (ICAC) Site, New York, New York
  - Cincinnati Children's Hospital Medical Center: Greater Cincinnati Pediatric Clinic Repository (GCPCR) and Mechanisms of Progression of Atopic Dermatitis to Asthma in Children (MPAACH) Site, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center: Inner City Asthma Consortium (ICAC) Site, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center: Outcome Measures in Eosinophilic Gastrointestinal Disorders Across the Ages (OMEGA) Site, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center:Cincinnati Childhood Allergy & Air Pollution Study (CCAAPS) Site, Cincinnati, Ohio
  - Vanderbilt University Medical Center: Infant Susceptibility to Pulmonary Infections and Asthma Following RSV Exposure Study (INSPIRE) Site, Nashville, Tennessee
  - University of Texas Southwestern Medical Center: Inner City Asthma Consortium (ICAC) Site, Dallas, Texas
  - University of Wisconsin Hospital and Clinics: Childhood Origins of Asthma (COAST) Site, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics: Wisconsin Infant Study Cohort (WISC) Site, Madison, Wisconsin

REFERENCES:
- [Derived] Moore CM, Secor EA, Everman JL, Fairbanks-Mahnke A, Jackson N, Pruesse E, Diener K, Morin A, Arbes SJ, Bacharier LB, Bendixsen CG, Calatroni A, Dupont WD, Furuta GT, Gebretsadik T, Gruchalla RS, Gupta RS, Khurana Hershey GK, Kattan M, Liu AH, Lussier SJ, Murrison LB, Numata M, O'Connor GT, Rivera-Spoljaric K, Phipatanakul W, Rothenberg ME, Seroogy CM, Zoratti EM, Castina S, Jackson DJ, Camargo CA Jr, Johnson CC, Ethridge R, Ramratnam S, Stelzig L, Teach SJ, Togias AG, Fulkerson PC, Hartert TV, Seibold MA. The Common Cold Is Associated With Protection From SARS-CoV-2 Infections. J Infect Dis. 2025 Dec 20;232(6):e920-e930. doi: 10.1093/infdis/jiaf374. PMID 40795882
- [Derived] Fulkerson PC, Lussier SJ, Bendixsen CG, Castina SM, Gebretsadik T, Marlin JS, Russell PB, Seibold MA, Everman JL, Moore CM, Snyder BM, Thompson K, Tregoning GS, Wellford S, Arbes SJ, Bacharier LB, Calatroni A, Camargo CA Jr, Dupont WD, Furuta GT, Gruchalla RS, Gupta RS, Hershey GK, Jackson DJ, Johnson CC, Kattan M, Liu AH, Murrison L, O'Connor GT, Phipatanakul W, Rivera-Spoljaric K, Rothenberg ME, Seroogy CM, Teach SJ, Zoratti EM, Togias A, Hartert TV, Heros Study Team OBOT. Human Epidemiology and Response to SARS-CoV-2 (HEROS): objectives, design, and enrollment results of a 12-city remote observational surveillance study of households with children, using direct-to-participant methods. Am J Epidemiol. 2024 Oct 7;193(10):1329-1338. doi: 10.1093/aje/kwae077. PMID 38775275
- See also: National Institute of Allergy and Infectious — http://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation — http://www.niaid.nih.gov/about/dait

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 01May2022 through 17Dec2020. Children and teenagers who were participating in NIH-funded cohorts that focused on asthma and/or allergic disease were recruited. In addition to the cohort-participating child, enrollment required a household caregiver; an additional household child and adult could also be enrolled.
Pre-assignment Details: The study was performed remotely. Participants completed a registration form and questionnaires/surveys electronically. Participants did a web-based training that described sample collection and handling, teletraining, & were provided written instructions. Study staff were available by phone, text, or video conferencing.The 2 main groups of interest in this study were "Index Participants" (the cohort-participating child) & "All Participants Combined" (index participant and household contacts).
Groups:
- Index Participants: Index participants are participants who are part of National Institutes of Health-funded cohorts that focused on asthma and/or allergic disease. This group will be index participants who enrolled in the study by completing the date on the electronic registration form and who also contributed at least 1 nasal swab while on study. This group is a subset of the group "All Participants Combined".
- Non-Index Participants: A minimum of 2 family members (index participant and a caregiver) and a maximum of 4 total family members (additional caregiver and/or sibling) were enrolled per family. This group is all participants excluding the index participants.
Period: Overall Study
Arm/Group | Index Participants | Non-Index Participants
Started | 1387 (Index participants who were enrolled and contributed at least 1 nasal swab) | 2755 (All participants who were enrolled and contributed at least 1 nasal swab)
Completed | 1012 (Index participants who at least started the exit survey) | 2011 (Participants who at least started the exit survey)
Not Completed | 375 | 744
Not completed — Death | 1 | 2
Not completed — Lost to Follow-up | 203 | 380
Not completed — Withdrawal by Subject | 47 | 98
Not completed — Noncompliance with study procedure | 121 | 251
Not completed — Reimbursement not enough | 1 | 2
Not completed — Unforeseen family circumstances | 1 | 3
Not completed — Test too painful | 1 | 1
Not completed — Moved | 0 | 2
Not completed — Nonresponsive | 0 | 5

BASELINE CHARACTERISTICS:
Population: Participants who enrolled in the study by completing the date on the electronic registration form and who also contributed at least 1 nasal swab while on study.
Groups:
- Index Participants: Index participants are participants who are part of National Institutes of Health-funded cohorts that focused on asthma and/or allergic disease. This group will be index participants who enrolled in the study by completing the date on the electronic registration form and who also contributed at least 1 nasal swab while on study.
- Non-Index Participants: A minimum of 2 family members (index participant and a caregiver) and a maximum of 4 total family members (additional caregiver and/or sibling) were enrolled per family. This group is all participants except Index Participants who enrolled in the study by completing the date on the electronic registration form and who also contributed at least 1 nasal swab while on study.
- Total: Total of all reporting groups
Arm/Group | Index Participants | Non-Index Participants | Total
Number analyzed (Participants) | 1387 | 2755 | 4142
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.3 (4.9) | 32.3 (15.8) | 25.0 (16.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 647 | 1756 | 2403
  Male | 734 | 993 | 1727
  Intersex | 1 | 3 | 4
  Unknown or Not Reported | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 174 | 302 | 476
  Not Hispanic or Latino | 1184 | 2406 | 3590
  Unknown or Not Reported | 29 | 47 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 20 | 30
  Asian | 23 | 55 | 78
  Native Hawaiian or Other Pacific Islander | 4 | 3 | 7
  Black or African American | 320 | 563 | 883
  White | 851 | 1854 | 2705
  More than one race | 86 | 83 | 169
  Unknown or Not Reported | 93 | 177 | 270
Region of Enrollment [Number; unit: participants]
  United States | 1387 | 2755 | 4142
Asthma [Count of Participants; unit: Participants] — Participants who reported asthma on the baseline survey
  Participants
    Yes | 528 | 622 | 1150
    No | 859 | 2133 | 2992
Food Allergies [Count of Participants; unit: Participants] — Participants who reported food allergies on the baseline survey
  Participants
    Yes | 343 | 306 | 649
    No | 1044 | 2449 | 3493
Eczema [Count of Participants; unit: Participants] — Participants who reported eczema (atopic dermatitis) on the baseline survey
  Participants
    Yes | 386 | 336 | 722
    No | 1001 | 2419 | 3420
Allergies (hay fever, rhinitis) [Count of Participants; unit: Participants] — Participants who reported allergies (hay fever, rhinitis) on the baseline survey
  Participants
    Yes | 685 | 1207 | 1892
    No | 702 | 1548 | 2250

OUTCOME MEASURES:

1. Primary Outcome: Number of Index Participants and Their Household Contacts With SARS-CoV-2 RNA Detection in Nasal Samples Over the Study/Surveillance Period
Description: Nasal samples were analyzed to determine whether a participant ever tested positive for SARS-CoV-2 or not over the course of the study. Kaplan-Meier was used to estimate survival probabilities at timepoints throughout the study. Participants were censored if they did not test positive for SARS-CoV-2 by the end of follow-up. The last positive nasal swab occurred at day 212.
Time Frame: Baseline through end of study (24 or 28 weeks, depending on if a participant agreed to do the extension)
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percent surviving using Kaplan-Meier
Groups:
- All Participants Combined: A minimum of 2 family members (index participant and a caregiver) and a maximum of 4 total family members (additional caregiver and/or sibling) were enrolled per family. This group is all participants who enrolled in the study by completing the date on the electronic registration form and who also contributed at least 1 nasal swab while on study.
Arm/Group | Index Participants | Non-Index Participants | All Participants Combined
Number analyzed (Participants) | 1387 | 2755 | 4142
Percent surviving using Kaplan-Meier
  30 Days | 98.9 [98.4 to 99.1] | 99.2 [98.8 to 99.5] | 99.1 [98.8 to 99.4]
  60 Days | 98.0 [97.3 to 98.8] | 98.4 [97.9 to 98.9] | 98.3 [97.9 to 98.7]
  90 Days | 97.2 [96.3 to 98.1] | 97.7 [97.1 to 98.3] | 97.5 [97.0 to 98.0]
  120 Days | 95.8 [94.7 to 96.9] | 96.1 [95.3 to 96.9] | 96.0 [95.3 to 96.6]
  150 Days | 94.2 [92.9 to 95.6] | 94.3 [93.3 to 95.2] | 94.3 [93.5 to 95.1]
  180 Days | 90.5 [88.5 to 92.7] | 91.4 [90.1 to 92.7] | 91.1 [90.0 to 92.2]
  210 Days | 90.1 [87.9 to 92.4] | 88.4 [85.3 to 91.7] | 89.0 [86.8 to 91.3]
  212 Days | 90.1 [87.9 to 92.4] | 83.5 [77.5 to 89.9] | 85.7 [81.5 to 90.1]

2. Secondary Outcome: Percent of Index Participants and Their Household Contacts With Detectable SARS-CoV-2-Specific Antibodies in Serum Over the Study/Surveillance Period
Description: Included: Participants currently or in the past enrolled in NIH-funded studies who fulfill inclusion criteria (index participant) and their family/household contacts.
  Outcome definition: Detectable SARS-CoV-2-specific antibodies in serum biological specimen(s).
Time Frame: Up to Week 24
Reporting Status: Not Posted

3. Secondary Outcome: Number of Index Participants With SARS-CoV-2 Detection in Nasal Samples With Asthma and Other Atopic Disease Compared to Index Participants Without Atopic Disease Over the Study/Surveillance Period
Description: Index participants: Those currently or in the past enrolled in NIH-funded studies who fulfill inclusion criteria.
  Testing method: Positive test result(s) for SARS-CoV-2 RNA in nasal samples.
Time Frame: Up to Week 24
Reporting Status: Not Posted

4. Secondary Outcome: Percent of Index Participants With Asthma and Other Atopic Disease With Detectable SARS-CoV-2-Specific Antibodies in Serum Compared to Index Participants Without Atopic Disease Over the Study/Surveillance Period
Description: Index participants: Those currently or in the past enrolled in NIH-funded studies who fulfill inclusion criteria.
  Outcome definition: Detectable SARS-CoV-2-specific antibodies in serum biological specimen(s).
Time Frame: Through study completion, an average of 24 Weeks
Reporting Status: Not Posted

5. Secondary Outcome: Changes in the Nasal Transcriptome Associated With Detection of SARS-CoV-2 in Nasal Samples Among Index Participants and Their Household Contacts Over the Study/Surveillance Period
Description: Nasal samples of participants currently or previously enrolled in NIH-funded studies who fulfill inclusion criteria (index participant) and their family/household contacts that test positive for SARS-CoV-2, will undergo transcriptome analysis.
  Total RNA will be isolated for cDNA synthesis and amplification. Differential gene expression analysis be pursued.
Time Frame: Up to Week 24
Reporting Status: Not Posted

6. Secondary Outcome: Changes in the Nasal Transcriptome Associated With Detection of SARS-CoV-2 in Nasal Samples Among Index Participants With Asthma and Other Atopic Disease Compared to Index Participants Without Atopic Disease Over the Study/Surveillance Period
Description: Nasal samples of index participants that test positive for SARS-CoV-2 will be evaluated by transcriptome analysis. Differential gene expression analysis at different timepoints in the disease process will be analyzed.
  Definition of index participant(s): Prior and/or current NIH-funded clinical research study participant(s) who fulfill inclusion criteria.
Time Frame: Up to Week 24
Reporting Status: Not Posted

7. Secondary Outcome: Symptoms Associated With Detection of SARS-CoV-2 in Nasal Samples Among Index Participants and Their Household Contacts Over the Study/Surveillance Period
Description: An analysis of symptoms associated with positive SARS-CoV-2 RNA tests in nasal samples will be conducted.
  Included in analysis: Index participants and their household contacts.
Time Frame: Up to Week 24
Reporting Status: Not Posted

8. Secondary Outcome: Number of Index Participants With SARS-CoV-2 Detection in Nasal Samples Using Topical Steroids Compared to Index Participants That Are Not Using Topical Steroids Over the Study/Surveillance Period
Description: Index participants: Those currently or in the past enrolled in NIH-funded studies who fulfill inclusion criteria.
  Tests: Positive for SARS-CoV-2 RNA in nasal samples
Time Frame: Up to Week 24
Reporting Status: Not Posted

9. Secondary Outcome: Number of Index Participants With SARS-CoV-2 Detection in Nasal Samples Using Topical, Oral, or Inhaled Steroids Compared to Index Participants That Are Not Using Topical, Oral, or Inhaled Steroids During the Study/Surveillance Period
Description: as for outcome 8
Time Frame: Up to Week 24
Reporting Status: Not Posted

10. Secondary Outcome: Analysis of Factors, Baseline and Prior History, for Possible Association With the Cumulative Incidence of SARS-COV-2 Detection in Nasal Samples: Index Participants and Their Household Contacts Over the Study/Surveillance Period
Description: An exploratory analysis will be conducted for detection of possible associations, focusing on baseline demographic and environment factors and/or history of bronchiolitis prior history with the cumulative incidence of SARS-CoV-2 detection in nasal samples Test: Positive for SARS-CoV-2 RNA in nasal samples.
Time Frame: Baseline, Week 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of first procedure, which occurred at study week 2, until a participant completed the study, until 48 hours after he/she prematurely withdrew, or is withdrawn from the study. Participants were followed for 24 or 28 weeks, or until they withdrew.
Description: Adverse events (including SAEs) were discovered by interviewing the participants through specific questions that were incorporated in the study questionnaires. Adverse events were also discovered if a participant had an unsolicited complaint. The two main groups of interest in this study were "Index Participants" (the cohort-participating child) and "All Participants Combined" (index participant and household contacts).
Arm/Group | Index Participants | Non-Index Participants
All-Cause Mortality (participants affected / at risk) | 0/1387 | 0/2755
Serious Adverse Events (participants affected / at risk) | 0/1387 | 0/2755
Other Adverse Events (participants affected / at risk) | 14/1387 | 4/2755
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Index Participants (N=1387) | Non-Index Participants (N=2755)
Vessel puncture site bruise (General disorders) | 3 (3) | 0 (0)
Vessel puncture site haemorrhage (General disorders) | 1 (1) | 0 (0)
Vessel puncture site hypoaesthesia (General disorders) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 1 (1) | 1 (1)
Vessel puncture site rash (General disorders) | 1 (1) | 0 (0)
Vessel puncture site swelling (General disorders) | 2 (2) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
34.4% of nasal collections were missed during the study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2020-09-02): https://cdn.clinicaltrials.gov/large-docs/61/NCT04375761/Prot_SAP_003.pdf
  • Informed Consent Form: Final ICF (2020-04-30): https://cdn.clinicaltrials.gov/large-docs/61/NCT04375761/ICF_001.pdf
  • Informed Consent Form: Adjustment ICF (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/61/NCT04375761/ICF_002.pdf